CLINICAL TRIAL: NCT00153556
Title: A Demonstration Project for the Elimination of Haemophilus Influenzae Type B in Three Rural Alaska Native Villages
Brief Title: Study to Eliminate Hib Carriage in Rural Alaska Native Villages
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: CDC-Arctic Investigations Program (Unknown); Alaska Native Tribal Health Consortium (Other); Yukon Kuskokwim Health Corporation (Other); Alaska State Public Health Laboratories (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-2961
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Haemophilus Influenzae Type B; Carrier State
Keywords: Haemophilus influenza type B; Carrier state; Bacterial Vaccines; Anti-PRP antibody; Antibody avidity; Serum bacteriocidal antibody; American Indians/Alaska Natives; Case control study; Adult vaccines
MeSH Terms: conditions — Haemophilus Infections

INTERVENTIONS:
Biological: Hib conjugate vaccine (HbOC, Wyeth Vaccines)

SUMMARY:
Hib disease rates in rural Alaska before introduction of HIb conjugate vaccine were among the highest in the world. Since vaccine introduction, rates have fallen by 90% but the disease has not been eliminated. This study is designed to test one possible means of eliminating Hib carriage and thus to eliminate person to person transmission and invasive disease.

The objective of this study is to evaluate the effectiveness of community-wide use of Hib conjugate vaccine for eliminating oropharyngeal Hib carriage in rural Alaska villages.

Secondary objectives include:

* Determine risk factors for Hib OP carriage including demographic characteristics, and immunologic characteristics (antibody level and function). This will be accomplished through a case-control study described below.
* Measure antibody response to Hib conjugate vaccine among adults who have not previously received Hib vaccine. This will be accomplished through a cohort study of participating adults in the vaccine intervention communities.

DETAILED DESCRIPTION:
This was a pilot intervention to assess the feasibility of using Hib conjugate vaccine to eliminate Hib carriage in rural Alaska villages, with three villages to serve as a comparison group. WE performed community-wide surveys of Hib carriage by recruiting volunteers for throat cultures to establish a baseline rate of Hib carriage for each community. Then Hib carriers were offered chemoprophylaxis to clear Hib from their throats. In the vaccine intervention communities, a single dose of Hib conjugate vaccine was offered to persons of all ages. This was followed by a second community-wide Hib carriage survey after one year to assess the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All village residents are eligible for Hib colonization survey
* All residents of selected villages eligible for vaccine study except as noted below.

Exclusion Criteria:

* For receipt of vaccine:
* history of allergic reaction to Hib vaccine or components
* Age < 24 months and not due for Hib vaccine according to childhood immunization schedule
* Age > 24 months and have received HIb vaccine within past year
* Pregnant

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3200
Dates: Start 2001-09; Study Completion 2003-11

PRIMARY OUTCOMES:
Change in community-wide oropharyngeal Hib colonization one year after administration of a single dose of Hib vaccine to all willing community members in 3 villages vs. change in HIb colonization in 3 village where Hib vaccine was used routinely

SECONDARY OUTCOMES:
- Safety of HIb vaccine given to adults
- Anti-PRP antibody/ avidity/ serum bacteriocidal activity among adult vaccine recipients, Hib colonized persons and age-matched controls
- Risk factors for Hib colonization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Hennessy, MD,MPH, Principal Investigator — Centers for Disease Control and Prevention-Arctic Investigations Program
Locations (1):
- CDC Arctic Investigations Program, Anchorage, Alaska, United States